CLINICAL TRIAL: NCT04517643
Title: Feasibility of a Personalized Dosimetry-based Treatment Planning for Radioembolization in the Treatment of Unresectable Colorectal Metastases in Liver
Brief Title: TheraSphere® For Treatment of Metastases in Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J2006; National Institute Of Health (Other Grant/Funding Number: HHSN267152N0911701090C3070C047)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: To investigate whether the dose predicted by pre-therapy 99mTc MAA SPECT predicts the dose to the liver from the 90Y microspheres as assessed by post-therapy 90Y SPECT/CT or PET/CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therasphere Therapy (Experimental): All participants will receive the Therasphere Therapy.
  Interventions: Other: Therasphere Therapy

INTERVENTIONS:
Other: Therasphere Therapy — TheraSphere is a radiotherapy treatment for primary and secondary liver neoplasia. This is an imaging study that will examine 3-5 patients who have been treated for metastatic colorectal cancer in the liver using TheraSphere®. Participation in the study involves an additional post-treatment SPECT/CT or PET/CT scan at (0-6) hours.

SUMMARY:
To investigate whether the dose predicted by pre-therapy 99mTc MAA SPECT predicts the dose to the liver from the 90Y microspheres as assessed by post-therapy 90Y SPECT/CT or positron emission tomography (PET)/CT.

DETAILED DESCRIPTION:
This study will acquire imaging information from 3-5 patients that will demonstrate feasibility of future implementation of personal dosimetry-based treatment planning for Trans-arterial Radio-embolization (TARE).

TARE therapy of liver neoplasia using 90Y-theraspheres has a long history. The device is FDA approved for the treatment of hepatocellular carcinoma, but has been used extensively for treatment of secondary liver neoplasia, including metastatic colorectal lesions under Humanitarian Device Exemption protocols such as this one.

As a targeted radioactive therapy, the current TARE implementation suffers from a lack of efficiency characteristic of radiopharmaceutical therapy (RPT) in general; namely, that the activity determined to treat the patient is not optimized according to normal organ tolerated absorbed dose and tumor efficacy thresholds. The amount of activity to be administered is determined from volumetrics established from associated imaging, either MRI or X-ray CT, where the total volume of irradiated tissue is considered as irrigated by the artery selected for administration, including both tumor and normal organ tissue. From this volume determination, the activity necessary to deliver an average pre-determined safe absorbed dose (120 Gy) to the entire irradiated region is calculated and administered.

In RPT, in the theranostic paradigm, a pre-therapeutic, or surrogate, quantity of activity is administered to the patient; 3D imaging (SPECT/CT or PET/CT) is then acquired at several time points and the individual patient's pharmacokinetics are determined, the normal organ and tumor dosimetry are performed and the optimal administered activity calculated that will deliver safe and efficacious treatment for the individual patient is determined, generally limited by the normal organ at risk maximum tolerated dose.

TARE presents a number of unique characteristics that enable a simpler version of this approach than is typical for most RPT. The method of administration means that only the normal liver and lungs need to be considered as potential organs at risk as the microspheres embolize and do not circulate systemically; the lack of associated photons in the 90Y decay chain means that a simple activity-to-dose-rate conversion can be used; the embolization means that only a single imaging time point is necessary as there is no redistribution of activity over time and the dose rate is converted to absorbed dose using the physical decay parameters of 90Y. These natural simplifications are already exploited in the current volumetric paradigm, where a 99mTc-macro albumin aggregate (MAA) surrogate and planar imaging are used to determine the fraction of total activity that is shunted to the lung and where a derived conversion factor is used to convert activity to absorbed dose.

The technical complication in TARE is that the surrogate (99mTc-MAA) has a different nature from the therapeutic device (90Y-theraspheres), and thus the reliability of the predictive quality of the surrogate is disputed. However, with precise and advanced imaging reconstruction and dosimetry the investigators have shown the ability to accurately and precisely predict normal liver and tumor average 90Y-therasphere uptake and absorbed dose from 99mTc-MAA.

This protocol seeks to acquire the imaging information from 3-5 patients that will demonstrate feasibility of future implementation of personal dosimetry-based treatment planning for TARE. In addition to the clinical standard of care assessments: 1. a single SPECT/CT instead of the current planar image will be acquired of the surrogate 99mTc-MAA; 2. An additional single 3D image (either SPECT/CT or PET/CT, depending on machine availability) will be acquired up to 6 hours post-administration of the therapeutic 90Y-microspheres for comparison. Informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* The Diagnosis of metastatic colorectal cancer to the liver
* Patients with a diagnosis of metastatic colorectal cancer to the liver
* Liver metastases are unresectable
* Tumors are hypervascular based on visual estimation by the Investigator
* Target tumors are measurable using standard imaging techniques
* Performance Status Score 0 - 2
* Age ≥18 years
* Life expectancy ≥3 months
* >4 weeks since prior radiation, surgery or chemotherapy
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines
* At least one month has elapsed since most recent prior cancer therapy with the following exception:
* Patient is willing to participate in the study and has signed the study informed consent

Exclusion Criteria:

Patients may not be treated with TheraSphere® if patients have any of the following exclusions:

* Any pre-treatment laboratory findings within 15 days of treatment demonstrating liver dysfunction:
* Blood test result levels outside of the normal range
* Any history of hepatic encephalopathy
* Any contraindications to angiography and hepatic artery catheterization such as:
* History of severe allergy or intolerance to any contrast media, narcotics, sedatives or atropine that cannot be corrected or premedicated
* Bleeding diathesis, not correctable by usual forms of therapy
* Severe peripheral vascular disease that would preclude catheterization.
* Evidence of pulmonary insufficiency
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Co-morbid disease or condition that would preclude safe delivery of TheraSphere® treatment or, in the judgment of the physician, place the patient at undue risk
* Pregnancy
* Special Categories of Patients: Not applicable
* Research in Mentally Disabled People: No. All participants or legal guardians will be fully able to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hobbs, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therasphere Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Therasphere Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white/caucasian | 3
  black/african american | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
met enrollment criteria as per protocol [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Met the Criterion That the Dose Estimated With Tc-99m MAA SPECT Was Within 15% of the Dose Estimated From Y-90 SPECT
Description: Change in dose estimates of radioactivity from Therasphere treatment to liver tumor target, measured in Gray, will be compared at pre-treatment and up to 6 hours post-treatment.
  Reported as number of patients that met the criterion that the dose estimated with Tc-99m MAA SPECT was within 15% of the dose estimated from Y-90 SPECT
Time Frame: Pre-Treatment and up to 6 hours Post-Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Therasphere Therapy
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: During SPECT/CT scan
Description: This study is unique in that it only involves one image (a spect scan) that occurs after a clinical procedure that involves the patient receiving a treatment with Therasphere.
  Regarding the scan itself, there were no associated AEs or deviations.
Arm/Group | Therasphere Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT04517643/Prot_SAP_000.pdf